CLINICAL TRIAL: NCT01169129
Title: Surgery and Whole Brain Radiotherapy Versus Whole Brain Radiotherapy and Radiosurgery for 1-3 Resectable Brain Metastases: Phase III Prospective Pilot Study
Brief Title: Surgery and Whole Brain Radiotherapy (RT) Versus Whole Brain Radiotherapy (RT) and Radiosurgery for 1-3 Resectable Brain Metastases
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3602010
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastases; Cancer
Keywords: brain metastases; radiosurgery; neurosurgery; surgery; radiotherapy; resectable brain metastases
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Brain Neoplasms | interventions — Surgical Procedures, Operative; Neurosurgical Procedures; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery+whole-brain irradiation (Active Comparator): brain metastases is resected and the patient is submitted to whole-brain irradiation
  Interventions: Other: surgery
- whole-brain irradiation+radiosurgery (Active Comparator): patients will be submitted to whole-brain irradiation and after, they will be submitted to radiosurgery.
  Interventions: Radiation: radiosurgery

INTERVENTIONS:
Other: surgery — resection of brain metastases
  Other Names: neurosurgery
  Arms: surgery+whole-brain irradiation
Radiation: radiosurgery — radiosurgery to brain metastases
  Other Names: stereotactic radiosurgery
  Arms: whole-brain irradiation+radiosurgery

SUMMARY:
Patients in good general condition with resectable brain metastases, looks better with more intense treatment of metastases. This local treatment has been accomplished with surgery or radiosurgery. However, there are no randomized studies comparing these two types of treatment. The purpose of this study is to make this.

DETAILED DESCRIPTION:
Patients in good general condition with resectable 1-3 brain metastases will be randomized to surgery and whole brain radiotherapy and whole brain radiotherapy and radiosurgery. Initially we will evaluate the feasibility of carrying out the study with 15 patients in each arm, and after, we will follow with the primary end-point of comparing the toxicity of the exclusively radiotherapy arm with complications of the surgical arm. As a secondary end-point, we will evaluate local recurrence-free survival, overall survival, distance cerebral relapse-free survival (metachronous brain metastasis), free of neurological progression survival, free of neurological death survival, free of dependent life (another person)survival , steroid-free survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology of primary tumors: all but primary small cell cancer, germ cell tumors, leukemia, lymphoma, or primary central nervous system.
* Primary-site: controlled, meaning operated and / or irradiated; without detectable local tumor activity
* Lack of extra-cranial metastases
* Absence of prior brain irradiation
* Number of brain metastases: 1-3
* Location of brain metastases: brain regions eligible for surgery (non-eloquent areas) and RC (metastases with largest diameter ≤ 3 cm, volume <15 mL, and> 5 mm from the optic chiasm, optic nerves, thalamus, hypothalamus, basal ganglia base, optic tract, optic radiation, midbrain, pons, medulla, corpus callosum, internal capsule, hippocampus and amygdala, and <10 ml of brain tissue receiving ≥ 12 Gy).
* Metastasis-that does not cause significant mass effect and hydrocephalus or herniation requiring urgent surgical intervention
* Second uncontrolled primary tumor site: none, except non-melanoma skin cancer
* Absence of comorbid conditions that prevents surgery for resection of brain metastases
* Absence of connective tissue disease such as lupus erythematosus or scleroderma
* Patients in chemotherapy need to have their chemotherapy treatment suspended.
* Patients must consent to be followed by clinical staff of the Barretos Cancer Hospital (HCB).
* KPS: ≥ 70%
* Neutrophils ≥ 1800 cells / mL until 14 days prior to study entry
* Platelets ≥ 100,000 cells / mL until 14 days prior to study entry
* Hemoglobin ≥ 10 g / dL 14 days prior to entering the study (transfusion is allowed to achieve required concentration)
* Creatinine ≤ 1.7 mg / dL 14 days prior to study entry
* BUN ≤ 30 mg / dL 14 days prior to entry on study
* Bilirubin ≤ 2 mg / dL 14 days prior to study entry
* TGO/TGP Up to three times normal on examination until 14 days prior to study entry Prothrombin time-INR <1.4 at examination until 14 days prior to study entry
* Systolic pressure ≤ 160 mm Hg and diastolic pressure ≤ 90 mm Hg at examination until 14 days prior to study entry Electrocardiogram-without acute myocardial infarction in examination until 14 days prior to study entry
* No active bleeding or pathological condition that entails high risk of bleeding
* Negative pregnancy test at least 14 days prior to study entry
* Informed Consent: The patient will be informed of the investigational nature of treatment and only enter the study after agreeing to participate in the study signed a consent form that informs the side effects and possible benefits and potential of both modalities treatment.

Exclusion Criteria:

* Metastasis in the posterior fossa, because this patient will be operated.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
feasibility | 1 year
  One year after the start of patient recruitment, the study will be analyzed for feasibility and, if feasible, we will pursue the study with primary end-point of comparing the toxicity of exclusive radiation therapy arm with the surgical arm.

SECONDARY OUTCOMES:
complications and toxicity | 1 year
  One year after the start of patient recruitment, the study will be analyzed for toxicity of the radiotherapy arm versus the arm surgical complications, and if compatible, will continue the study until 70 patients in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Nakamura, MD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil